CLINICAL TRIAL: NCT00964808
Title: Norspan Versus Oxycontin as Postoperative Painkiller to Proximal Extracapsular Fractures of the Femur
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Vejle Hospital (Other)
Collaborators: Norpharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EudraCT2009-010539-41
Record Dates: First submitted 2009-08-24; First posted 2009-08-25 (Estimated); Last update posted 2014-12-08 (Estimated); Status verified 2014-12

CONDITIONS: Pain, Postoperative
Keywords: Hip fractures; Treatment Outcome; Painkiller
MeSH Terms: conditions — Pain, Postoperative; Hip Fractures | interventions — Buprenorphine; Oxycodone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Buprenorphine (Experimental): Double dummy; Group A: Active Buprenorphine and placebo oxycodone
  Interventions: Drug: Buprenorphine
- Oxycodone (Experimental): Double Dummy:
  Group B: Placebo Buprenorphine and Active Oxycodone
  Interventions: Drug: Oxycodone

INTERVENTIONS:
Drug: Buprenorphine — Start: Day 0 (T=0), 10 micrograms/t until the day of discharge from the Hospital. New plaster at T= 7 days.
  Other Names: Norspan
  Arms: Buprenorphine
Drug: Oxycodone — Start: 10 hours (+/- 2 hours) after the operation. Dosage: 10 mg * 2 pr. day until time to discharge from the Hospital or latest at day 12.
  Other Names: Oxycontin
  Arms: Oxycodone

SUMMARY:
Effective treatment of pain after hip fractures is very important but difficult. It is often an old patient who has many adverse effects with the use of morphine.

This is a randomized pilot study where the investigators want to compare Norspan plaster to Oxycontin tablets to patients with particular kind of hip fractures. The investigators will evaluate mobilization, pain, use of rescue medicine, adverse effects and length of stay. No clinical study about the effect of Norspan as acute painkiller has never been done before. Can the investigators get the patients mobilized earlier with less adverse effects?

ELIGIBILITY:
Inclusion Criteria:

* Males and females age 18 years or more
* X-ray confirming basicervical, pertrochanteric or subtrochanteric femur fracture and planning operation with DHS or PFN.
* Subjects must have 7 or more points in the Hindsøes test.

Exclusion Criteria:

* Subjects where spinal anaesthesia cannot be applied.
* Subject in Plavix® treatment seven days before admission to the hospital.
* Subjects with extracapsular hip fracture due to bone metastasis.
* Subjects with a BMI over 30.
* Subjects under 45 kg.
* Subjects who are currently taking monoamine oxidase inhibitors (MAOIs) or have taken MAOIs within 2 weeks prior admission to the hospital.
* Substance or alcohol abuse, or subjects who, in the opinion of the investigator have demonstrated addictive or substance abuse behavior.
* Untreated depression or other psychiatric disorder in such a way that participation in the study may in the opinion of the investigator pos an unacceptable risk to the subject.
* Dermatological disorder at any relevant patch application site.
* Any contraindications listed in the Summary of Product Characteristics for Norspan®, OxyNorm® and OxyContin®.
* Patient does not tolerate oxynorm.
* User of wheelchair.
* Daily use of morphine before hospitalization.
* More than one fracture. Patients with myasthenia gravis. Patients with severe respiratory function. Patients know need re-operation women of childbearing potential must have a negative pregnancy test and be non-lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-09; Primary Completion 2013-05 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Mobilization measured daily using Cumulated Ambulation Score. | 12 days

SECONDARY OUTCOMES:
Pain intensity measured daily on a verbal rating scale | 12 days
Adverse effects | 12 days + 14 days
Opioid consumption. | 12 days
Length of stay in Hospital | Untill discharge

CONTACTS AND LOCATIONS:
Overall Officials: Per Kjaersgaard-Andersen, MD, Study Director — Orthopaedic Department, Vejle Hospital, Denmark
Locations (1):
- Orthopaedic Department, Vejle, Denmark